CLINICAL TRIAL: NCT06492590
Title: Assessing a Multicomponent Intervention to Improve Quality of Life in Individuals With Long COVID-19 (COVIDL/MIQoL): A Randomized Controlled Trial
Brief Title: Long COVID-19 Intervention (COVIDL/MIQoL)
Acronym: COVIDL/MIQoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Maria Llistosella, Principal Investigator, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PT-082023-EP HUB
Record Dates: First submitted 2024-07-08; First posted 2024-07-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Long COVID-19
Keywords: Physical Rehabilitation; Psychological Intervention; Randomized Controlled Trial; Long COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: This study is a Randomized controlled trial with parallel arms. Participants will be randomly allocated either to an intervention group or control by the external researcher using computer-generated random numbers
Masking Description: No-blinded participant and personnel (research team).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A multicomponent intervention: The psycho-education will consist of 9 sessions of 90 minutes, one per week, in groups of a maximum of 16 participants.The topics that will be covered during the sessions with a specialized therapist will be: (1) education in neuroscience of the symptomatology of the Long COVID; (2) Mindfulness; (3) Cognitive-Behavioral Therapy; and (4) Strategies of self-healing. Physical rehabilitation will consist of 9 sessions of 60 minutes, one per week, in groups of a maximum of 16 participants, conducted by an expert physiotherapist. Each session will work on the following 4 blocks in a progressive approach: (1) warm-up and aerobic exercises (25 minutes); (2) functional and muscle strengthening exercises (10 minutes); (3) Proprioception exercises (10 minutes); and (4) breathing exercises (10 minutes). Answering the assessment questionnaires pre, post and 24 weeks of intervention follow-up
  Interventions: Behavioral: Multicomponent intervention
- Control group (No Intervention): Participants in the control group will complete the same research questionnaires as the intervention group and for the same period.
  Participants in the control group will be placed on a waiting list for the intervention once its efficacy has been demonstrated.

INTERVENTIONS:
Behavioral: Multicomponent intervention — Multicomponent intervention based on psycho-education and physical rehabilitation.
  Other Names: COVID-L/MIQoLI
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of a multicomponent intervention in individuals with Long COVID. The main questions it aims to answer are:

* Does the intervention increase quality of life, mental well-being, resilience, and physical condition in individuals with Long COVID?
* Does the intervention decrease anxiety, depressed mood, and fatigue in individuals with Long COVID? The researchers will compare the multicomponent intervention with a control (non-intervention) group.

Participants will:

• Participate in a multicomponent intervention for 9 weeks (2 sessions each week, one of psycho-education and one of physical rehabilitation).

DETAILED DESCRIPTION:
Background The persistence of symptoms after acute SARS-CoV-2 infection, known as Long COVID, has emerged as a wide-ranging public health challenge. This condition, characterised by a wide range of physical and psychological symptoms that persist months after initial recovery, significantly affects patients' quality of life.

To our knowledge, in the Primary Health Care setting, there are few published clinical trials of multicomponent interventions involving psycho-educational and physical rehabilitation activities to improve quality of life of individuals with Long COVID. Therefore, the purpose of this trial is to assess the effectiveness of an innovative multicomponent intervention, which includes psycho-education and physical rehabilitation and which is in line with the complex needs of individuals with Long COVID.

The investigators hypothesize that participants with Long COVID, who receive the multicomponent intervention (psycho-education and physical rehabilitation), will increase their quality of life, mental well-being, resilience, and physical condition; and decreased anxiety, depressed mood, and fatigue compared to the control group.

Method The study is a Randomized Controlled Trial (RCT). Participants will sign an agreement to participate in the study and will be randomly allocated in control and intervention groups by external researcher using a computer-generated random number.

The intervention will be carried out during January (2025)- September (2025). Participants will follow a specific training consisting of 18 sessions: 9 sessions (psycho-education) of 90 minutes, one per week conducted by specialized therapist; and 9 sessions (physical rehabilitation) of 60 minutes, one per week, conducted by an expert physiotherapist.

The data collection will start in January 2025 and will finish in September 2025. Data will be collected at baseline before the intervention (T0), after 9 weeks post-intervention (T1) and 24 weeks follow-up (T2).

The assessment of the effectiveness of the intervention will be carried out using the psychometric scale EuroQol5D-5L (as the primary outcome) which will allow the investigators to determine changes in quality of live.

Using SD of the primary outcome EuroQol5D-5L, minimum sample size was calculated to be 34 participants in each group, using GRANMO (https://www.imim.es/ofertadeserveis/software-public/granmo/). A follow-up loss rate of 10% was estimated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Long COVID-19
* Present discomfort with the situation
* Individuals aged 18 to 75
* Sign the informed consent form

Exclusion Criteria:

* Severe sensory deficits
* Physical illnesses that do not allow attendance at the sessions
* Severe mental disorders that make participation in groups inadvisable
* Travel, surgery, or other event that does not allow at least 80% of the sessions
* No comprehension of the language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male, female, non-binary
Enrollment: 74 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Improved quality of life | Baseline (T0), post-intervention (9 weeks) (T1), and 24 weeks follow-up (T2)
  Changes in level of quality of life using the EuroQol 5D-5L scale (EQ-5D-5L). Values range from 0 to 1 (full health). Higher scores, better outcome

SECONDARY OUTCOMES:
Improve well-being | Baseline (T0), post-intervention (9 weeks) (T1), and 24 weeks follow-up (T2)
  Changes in level of well-being using the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). Values range from 14 to 70 . Higher scores, better outcome
Decreased anxiety and depression | Baseline (T0), post-intervention (9 weeks) (T1), and 24 weeks follow-up (T2)
  Changes in level of anxiety and depression using the Hospital Anxiety and Depression Scale (HADS). Anxiety values range from 0 to 15 . Higher scores, worse outcome. Depression values range from 0 to 12. Higher scores, worse outcome
Increased resilience | Baseline (T0), post-intervention (9 weeks) (T1), and 24 weeks follow-up (T2)
  Changes in level of resilience using the Connor-Davidson Resilience Scale (CD-RISC). Values range from 0 to 40 . Higher scores, better outcome
Improve physical activity | Baseline (T0), post-intervention (9 weeks) (T1), and 24 weeks follow-up (T2)
  Changes in level of physical activity using the International Physical Activity Questionnaire (IPAQ). In each category a maximum of 21 hours of activity are permitted a week (3 hours X 7 days) To calculate MET minutes a week multiply the MET value given (r walking = 3.3, moderate activity = 4, vigorous activity = 8) by the minutes the activity was carried out and again by the number of days that that activity was undertaken. Higher scores, better outcome
Decreased fatigue | Baseline (T0), post-intervention (9 weeks) (T1), and 24 weeks follow-up (T2)
  Changes in level of fatigue scale using the Chalder Fatigue Scale (CFS). Values range from 0 to 42 . Higher scores, worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Llistosella, PhD, Principal Investigator — Primary Health Care, Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Hernandez G, Garin O, Pardo Y, Vilagut G, Pont A, Suarez M, Neira M, Rajmil L, Gorostiza I, Ramallo-Farina Y, Cabases J, Alonso J, Ferrer M. Validity of the EQ-5D-5L and reference norms for the Spanish population. Qual Life Res. 2018 Sep;27(9):2337-2348. doi: 10.1007/s11136-018-1877-5. Epub 2018 May 16. PMID 29767329
- [Background] Castellvi P, Forero CG, Codony M, Vilagut G, Brugulat P, Medina A, Gabilondo A, Mompart A, Colom J, Tresserras R, Ferrer M, Stewart-Brown S, Alonso J. The Spanish version of the Warwick-Edinburgh mental well-being scale (WEMWBS) is valid for use in the general population. Qual Life Res. 2014 Apr;23(3):857-68. doi: 10.1007/s11136-013-0513-7. Epub 2013 Sep 5. PMID 24005886
- [Background] Herrero MJ, Blanch J, Peri JM, De Pablo J, Pintor L, Bulbena A. A validation study of the hospital anxiety and depression scale (HADS) in a Spanish population. Gen Hosp Psychiatry. 2003 Jul-Aug;25(4):277-83. doi: 10.1016/s0163-8343(03)00043-4. PMID 12850660
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Roman Vinas B, Ribas Barba L, Ngo J, Serra Majem L. [Validity of the international physical activity questionnaire in the Catalan population (Spain)]. Gac Sanit. 2013 May-Jun;27(3):254-7. doi: 10.1016/j.gaceta.2012.05.013. Epub 2012 Oct 24. Spanish. PMID 23103093
- [Background] Jackson C. The Chalder Fatigue Scale (CFQ 11). Occup Med (Lond). 2015 Jan;65(1):86. doi: 10.1093/occmed/kqu168. No abstract available. PMID 25559796
- [Background] Nury Nusdwinuringtyas, Kevin Triangto, Idrus Alwi, Faisal Yunus. The Validity and Reliability of Six Minute Walk Test in a 15 Meter Track. Indones J Phys Med Rehabil. 2022;10(02).
- [Derived] Morera M, Arevalo A, Garriga C, Corral-Magana M, Garcia-Arque MC, Gragea-Nocete M, Perez Diaz C, Roca R, Llistosella M. Assessing a multicomponent intervention to improve quality of life in individuals with Long COVID (COVIDL/MIQoL): study protocol for a randomized controlled trial. Front Public Health. 2025 May 19;13:1604971. doi: 10.3389/fpubh.2025.1604971. eCollection 2025. PMID 40458104
- See also: Situació actual de la COVID-19 persistent a Catalunya. Càrrega estimada, recursos assistencials, experiències internacionals i àrees d'incertesa. Comitè Científic Assessor de la COVID-19 — https://salutpublica.gencat.cat/web/.content/minisite/aspcat/sobre_lagencia/comite_assessor_covid19/230120_Informe-Long-Covid-.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT06492590/Prot_SAP_000.pdf